CLINICAL TRIAL: NCT06494761
Title: The Effect of Multiple Doses of Zongertinib on the Single-dose Pharmacokinetics of Midazolam, Omeprazole and Repaglinide in Healthy Male Subjects (an Open-label, 2-period, Fixed-sequence Trial)
Brief Title: A Study in Healthy Men to Test Whether Zongertinib Affects How 3 Other Medicines (Midazolam, Omeprazole, and Repaglinide) Are Taken up and Processed by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0014; 2023-510263-35-00 (Registry Identifier: CTIS); U1111-1301-9035 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Omeprazole; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Repaglinide+Midazolam+Omeprazole (Reference)/ Zongertinib+Repaglinide+Midazolam+Omeprazole (Test) (Experimental): Reference (Repaglinide + Midazolam + Omeprazole)
  In the reference treatment period (Period 1), participants received 0.5 mg repaglinide tablet (Day 1, after ≥10 h fast; Reference Treatment 1). On Day 2, they received 1 mg midazolam (0.5 mL oral solution) with 20 mg omeprazole tablet under the same fasting conditions (Reference Treatment 2).
  Test (Zongertinib + Repaglinide + Midazolam + Omeprazole)
  In the test treatment period (Period 2), participants received multiple once-daily doses of 120 mg zongertinib from Day 1 to Day 15. A single 0.5 mg repaglinide tablet was co-administered on Day 1 (Test Treatment 1) and Day 14 (Test Treatment 3), and a single dose of the probe drug cocktail containing 1 mg midazolam (0.5 mL oral solution) and 20 mg omeprazole tablet was co-administered on Day 2 (Test Treatment 2) and Day 15 (Test Treatment 4).
  Interventions: Drug: zongertinib; Drug: midazolam; Drug: omeprazole; Drug: repaglinide

INTERVENTIONS:
Drug: zongertinib — Participants received 120 mg Zongertinib daily as two 60 mg tablets.
  Other Names: BI 1810631
Drug: midazolam — Participants received 1 mg Midazolam as 0.5 mL oral solution.
Drug: omeprazole — Participants received 20 mg Omeprazole.
Drug: repaglinide — Participants received a 0.5 mg Repaglinide.

SUMMARY:
The main objective of this trial is to assess the effect of multiple oral doses of zongertinib on the pharmacokinetics of midazolam, omeprazole and repaglinide.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-randomized, open-label, two-period, fixed-sequence trial evaluated the effect of multiple oral doses of zongertinib on the single-dose pharmacokinetics of midazolam, omeprazole, and repaglinide in healthy male subjects to assess potential drug-drug interactions.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Period 1 (Reference Period) (3 days)
Arm/Group | Repaglinide+Midazolam+Omeprazole (Reference)/ Zongertinib+Repaglinide+Midazolam+Omeprazole (Test)
Started (Started Trial Medication) | 16
Completed (Completed Trial Medication) | 16
Not Completed | 0
Period: Washout (3 days)
Arm/Group | Repaglinide+Midazolam+Omeprazole (Reference)/ Zongertinib+Repaglinide+Midazolam+Omeprazole (Test)
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2: (Test Period) (15 days)
Arm/Group | Repaglinide+Midazolam+Omeprazole (Reference)/ Zongertinib+Repaglinide+Midazolam+Omeprazole (Test)
Started (Started Trial Medication) | 16
Completed (Completed Trial Medication) | 14
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
Arm/Group | Repaglinide+Midazolam+Omeprazole (Reference)/ Zongertinib+Repaglinide+Midazolam+Omeprazole (Test)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] — Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
  Years | 35.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
  Participants
    Female | 0
    Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 16
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 16
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Repaglinide in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC₀-∞)
Description: The area under the concentration-time curve of repaglinide in plasma over the time interval from 0 extrapolated to infinity ((AUC0-∞) is reported.
  Period 1 (Day 1): Up to 3 hours pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3-, 4-, 6-, and 24-hours post-dose. Period 2 (Day 1): Up to 3 hours pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3-, 4-, 6-, and 24-hours post-dose. Period 2 (Day 14): ≤15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 2.5, 3-, 4-,6-, and 24-hours post-dose.
Time Frame: Samples were collected on Day 1 (Period 1), Day 1 (Period 2), and Day 14 (Period 2). See endpoint description for the full sampling schedule
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Two subjects were discontinued by the investigator before Zongertinib administration on Day 2, leading to fewer subjects in Test Treatment 3 Arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours × picomoles per liter (h*pmol/L)
Groups:
- Repaglinide Alone (Reference Treatment 1): In the reference treatment period (Period 1), participants received a single oral dose of 0.5 mg repaglinide on Day 1 following an overnight fast of at least 10 hours.
- Repaglinide with a single dose of zongertinib (Test Treatment 1): In the test treatment period (Period 2), Day 1, participants received a single 0.5 mg dose of repaglinide coadministered with a single 120 mg dose of zongertinib (two 60 mg tablets) following an overnight fast of at least 10 hours.
- Repaglinide after multiple doses of zongertinib (Test Treatment 3): In the test treatment period (period 2), participants received 120 mg zongertinib (two 60 mg tablets) daily for 13 consecutive days. On Day 14, after 13 days of zongertinib administration, a single dose of 0.5 mg repaglinide tablet was coadministered with 120 mg zongertinib following an overnight fast of at least 10 hours.
Arm/Group | Repaglinide Alone (Reference Treatment 1) | Repaglinide with a single dose of zongertinib (Test Treatment 1) | Repaglinide after multiple doses of zongertinib (Test Treatment 3)
Number analyzed (Participants) | 16 | 16 | 14
Hours × picomoles per liter (h*pmol/L) | 28100 (58.0) | 31200 (49.2) | 37300 (48.7)
Statistical Analysis 1: Comparison: Repaglinide Alone (Reference Treatment 1) vs Repaglinide with a single dose of zongertinib (Test Treatment 1); The relative bioavailability of Repaglinide was assessed by comparing Repaglinide administered with a single dose of zongertinib (Test Treatment 1) to Repaglinide administered alone (Reference Treatment 1). The ratio of geometric means (Test/Reference) with 90% two-sided confidence intervals (CIs) was calculated. The log-transformed difference (log[T]-log[R]) was estimated using least squares means from ANOVA and then back-transformed to the original scale; Test type: Other; Ratios of adjusted geometric means [%] = 110.98, 90% CI 2-sided [96.90 to 127.10] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 22.1
Statistical Analysis 2: Comparison: Repaglinide Alone (Reference Treatment 1) vs Repaglinide after multiple doses of zongertinib (Test Treatment 3); The relative bioavailability of Repaglinide was assessed by comparing Repaglinide administered after multiple doses of zongertinib (Test Treatment 3) to Repaglinide administered alone (Reference Treatment 1). The ratio of geometric means (Test/Reference) with 90% two-sided confidence intervals (CIs) was calculated. The log-transformed difference (log[T]-log[R]) was estimated using least squares means from ANOVA and then back-transformed to the original scale; Test type: Other; Ratios of adjusted geometric means [%] = 130.10, 90% CI 2-sided [110.35 to 153.39] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 25.2

2. Primary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC₀-∞)
Description: The area under the concentration-time curve of midazolam in plasma over the time interval from 0 extrapolated to infinity ((AUC0-∞) is reported.
  Period 1 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 hours post-dose. Period 2 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 h post-dose. Period 2 (Day 15): 15 min pre-dose, and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 11, 12 hours post-dose.
Time Frame: Samples were collected on Day 2 (Period 1), Day 2 (Period 2), and Day 15 (Period 2). See endpoint description for the full sampling schedule
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Two subjects were discontinued by the investigator before Zongertinib administration on Day 2, leading to fewer subjects in Test Treatment Arm 2 and 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours × picomoles per liter (h*pmol/L)
Groups:
- Midazolam + Omeprazole (Reference Treatment 2): In the reference treatment period (Period 1), participants received a single oral dose of 1 mg Midazolam (0.5 mL oral solution) on Day 2, coadministered with a 20 mg Omeprazole tablet following an overnight fast of at least 10 hours.
- Midazolam + Omeprazole with a single dose of zongertinib (Test Treatment 2): In the test treatment period (Period 2), participants received 120 mg zongertinib (two 60 mg tablets) on Day 1. On Day 2, after one day of zongertinib pretreatment, participants were administered 1 mg, midazolam, coadministered with 20 mg omeprazole, and zongertinib following an overnight fast of at least 10 hours.
- Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4): In the test treatment period (Period 2), participants received 120 mg Zongertinib daily (two 60 mg tablets) for 14 consecutive days. On Day 15, after 14 days of zongertinib treatment, participants received 1 mg midazolam, coadministered with 20 mg omeprazole, and zongertinib following an overnight fast of at least 10 hours.
Arm/Group | Midazolam + Omeprazole (Reference Treatment 2) | Midazolam + Omeprazole with a single dose of zongertinib (Test Treatment 2) | Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4)
Number analyzed (Participants) | 16 | 14 | 14
Hours × picomoles per liter (h*pmol/L) | 41400 (33.5) | 44200 (37.3) | 43400 (27.9)
Statistical Analysis 1: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole with a single dose of zongertinib (Test Treatment 2); The relative bioavailability of midazolam was assessed by comparing Midazolam + Omeprazole with a single dose of zongertinib (Test Treatment 2) to Midazolam + Omeprazole (Reference Treatment 2). The ratio of geometric means (Test/Reference) with 90% two-sided confidence intervals (CIs) was calculated. The log-transformed difference (log[T]-log[R]) was estimated using least squares means from ANOVA and then back-transformed to the original scale; Test type: Other; Ratios of adjusted geometric means [%] = 107.80, 90% CI 2-sided [98.57 to 117.90] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 13.5
Statistical Analysis 2: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4); The relative bioavailability of midazolam was assessed by comparing Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4) to Midazolam + Omeprazole (Reference Treatment 2). The ratio of geometric means (Test/Reference) with 90% two-sided confidence intervals (CIs) was calculated. The log-transformed difference (log[T]-log[R]) was estimated using least squares means from ANOVA and then back-transformed to the original scale; Test type: Other; Ratios of adjusted geometric means [%] = 105.62, 90% CI 2-sided [95.41 to 116.93] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 15.4

3. Primary Outcome: Area Under the Concentration-time Curve of Omeprazole in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC₀-∞)
Description: The area under the concentration-time curve of omeprazole in plasma over the time interval from 0 extrapolated to infinity ((AUC0-∞) is reported.
  Period 1 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 hours post-dose. Period 2 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 h post-dose. Period 2 (Day 15): 15 min pre-dose, and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 11, 12 hours post-dose.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with evaluable results were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanogram per milliliter (h*ng/mL)
Groups:
- Midazolam + Omeprazole (Reference Treatment 2): In the reference treatment period (Period 1), participants received 1 mg midazolam (0.5 mL oral solution) coadministered with a 20 mg omeprazole tablet on Day 2 following an overnight fast of at least 10 hours.
- Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2): In the test treatment period (Period 2), participants received 120 mg zongertinib (two 60 mg tablets) on Day 1. On Day 2, after one day of zongertinib pretreatment, participants were administered 1 mg, midazolam, coadministered with 20 mg omeprazole, and zongertinib following an overnight fast of at least 10 hours.
Arm/Group | Midazolam + Omeprazole (Reference Treatment 2) | Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2) | Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4)
Number analyzed (Participants) | 10 | 10 | 9
hour * nanogram per milliliter (h*ng/mL) | 378 (69.7) | 359 (66.9) | 296 (60.2)
Statistical Analysis 1: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2); The relative bioavailability of omeprazole was assessed by comparing Midazolam + Omeprazole with a single dose of zongertinib (Test Treatment 2) to Midazolam + Omeprazole (Reference Treatment 2). The ratio of geometric means (Test/Reference) with 90% two-sided confidence intervals (CIs) was calculated. The log-transformed difference (log[T]-log[R]) was estimated using least squares means from ANOVA and then back-transformed to the original scale; Test type: Other; Ratios of adjusted geometric means [%] = 96.55, 90% CI 2-sided [75.96 to 122.72] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 24.5
Statistical Analysis 2: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4); The relative bioavailability of omeprazole was assessed by comparing Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4) to Midazolam + Omeprazole (Reference Treatment 2). The ratio of geometric means (Test/Reference) with 90% two-sided confidence intervals (CIs) was calculated. The log-transformed difference (log[T]-log[R]) was estimated using least squares means from ANOVA and then back-transformed to the original scale; Test type: Other; Ratios of adjusted geometric means [%] = 89.75, 90% CI 2-sided [61.86 to 130.20] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 39.6

4. Primary Outcome: Maximum Measured Concentration of Repaglinide in Plasma (Cmax)
Description: The maximum measured concentration of repaglinide in plasma is reported.
  Period 1 (Day 1): Up to 3 hours pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3-, 4-, 6-, and 24-hours post-dose. Period 2 (Day 1): Up to 3 hours pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3-, 4-, 6-, and 24-hours post-dose. Period 2 (Day 14): ≤15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 2.5, 3-, 4-,6-, and 24-hours post-dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles per liter (pmol/L)
Groups:
- Repaglinide with a single dose of zongertinib (Test Treatments 1): In the test treatment period (Period 2), Day 1, participants received a single 0.5 mg dose of repaglinide coadministered with a single 120 mg dose of zongertinib (two 60 mg tablets) following an overnight fast of at least 10 hours.
Arm/Group | Repaglinide Alone (Reference Treatment 1) | Repaglinide with a single dose of zongertinib (Test Treatments 1) | Repaglinide after multiple doses of zongertinib (Test Treatment 3)
Number analyzed (Participants) | 16 | 16 | 14
Picomoles per liter (pmol/L) | 20200 (52.6) | 23600 (40.9) | 29700 (36.8)
Statistical Analysis 1: Comparison: Repaglinide Alone (Reference Treatment 1) vs Repaglinide with a single dose of zongertinib (Test Treatments 1); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 117.07, 90% CI 2-sided [105.56 to 129.84] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 16.8
Statistical Analysis 2: Comparison: Repaglinide Alone (Reference Treatment 1) vs Repaglinide after multiple doses of zongertinib (Test Treatment 3); [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratios of adjusted geometric means [%] = 144.36, 90% CI 2-sided [123.53 to 168.71] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 23.9

5. Primary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax)
Description: The maximum measured concentration of midazolam in plasma is reported.
  Period 1 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 hours post-dose. Period 2 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 h post-dose. Period 2 (Day 15): 15 min pre-dose, and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 11, 12 hours post-dose.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles per liter (pmol/L)
Arm/Group | Midazolam + Omeprazole (Reference Treatment 2) | Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2) | Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4)
Number analyzed (Participants) | 16 | 14 | 14
Picomoles per liter (pmol/L) | 17700 (25.8) | 19700 (33.0) | 20800 (26.0)
Statistical Analysis 1: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 110.74, 90% CI 2-sided [100.92 to 121.52] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 14.1
Statistical Analysis 2: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4); [analysis description as in outcome 2, analysis 2]; Test type: Other; Ratios of adjusted geometric means [%] = 117.19, 90% CI 2-sided [108.30 to 126.81] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 11.9

6. Primary Outcome: Maximum Measured Concentration of Omeprazole in Plasma (Cmax)
Description: The maximum measured concentration of omeprazole in plasma is reported.
  Period 1 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 hours post-dose. Period 2 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 h post-dose. Period 2 (Day 15): 15 min pre-dose, and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 11, 12 hours post-dose.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Midazolam + Omeprazole (Reference Treatment 2) | Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2) | Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4)
Number analyzed (Participants) | 15 | 13 | 13
Nanograms per milliliter (ng/mL) | 165 (91.7) | 131 (78.3) | 101 (79.3)
Statistical Analysis 1: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2); [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 79.39, 90% CI 2-sided [49.90 to 126.30] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 77.6
Statistical Analysis 2: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4); [analysis description as in outcome 3, analysis 2]; Test type: Other; Ratios of adjusted geometric means [%] = 62.07, 90% CI 2-sided [44.69 to 86.20] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 49.1

7. Secondary Outcome: Area Under the Concentration-time Curve of Repaglinide in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: The area under the concentration-time curve of repaglinide in plasma over the time interval from 0 to the last quantifiable data poin is reported.
  Period 1 (Day 1): Up to 3 hours pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3-, 4-, 6-, and 24-hours post-dose. Period 2 (Day 1): Up to 3 hours pre-dose and at 15, 30, and 45 minutes, and 1, 1.5, 2, 2.5, 3-, 4-, 6-, and 24-hours post-dose. Period 2 (Day 14): ≤15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 2.5, 3-, 4-,6-, and 24-hours post-dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours × picomoles per liter (h*pmol/L)
Groups:
- Repaglinide after multiple doses of zongertinib (Test Treatment 3): In the test treatment period (period 2), participants received 120 mg zongertinib (two 60 mg tablets) daily for 13 consecutive days. On Day 14, following 13 days of zongertinib administration, a single dose of 0.5 mg repaglinide tablet was coadministered with 120 mg zongertinib following an overnight fast of at least 10 hours.
Arm/Group | Repaglinide Alone (Reference Treatment 1) | Repaglinide with a single dose of zongertinib (Test Treatments 1) | Repaglinide after multiple doses of zongertinib (Test Treatment 3)
Number analyzed (Participants) | 16 | 16 | 14
Hours × picomoles per liter (h*pmol/L) | 27700 (58.3) | 30700 (50.5) | 36700 (48.7)
Statistical Analysis 1: Comparison: Repaglinide Alone (Reference Treatment 1) vs Repaglinide with a single dose of zongertinib (Test Treatments 1); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 110.86, 90% CI 2-sided [96.58 to 127.24] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 22.5
Statistical Analysis 2: Comparison: Repaglinide Alone (Reference Treatment 1) vs Repaglinide after multiple doses of zongertinib (Test Treatment 3); [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratios of adjusted geometric means [%] = 129.80, 90% CI 2-sided [109.70 to 153.59] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 25.8

8. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: The area under the concentration-time curve of midazolam in plasma over the time interval from 0 to the last quantifiable data point is reported.
  Period 1 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 hours post-dose. Period 2 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 h post-dose. Period 2 (Day 15): 15 min pre-dose, and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 11, 12 hours post-dose.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours × picomoles per liter (h*pmol/L)
Arm/Group | Midazolam + Omeprazole (Reference Treatment 2) | Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2) | Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4)
Number analyzed (Participants) | 16 | 14 | 14
Hours × picomoles per liter (h*pmol/L) | 39600 (33.6) | 42700 (38.1) | 41700 (27.7)
Statistical Analysis 1: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2); [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 108.61, 90% CI 2-sided [98.79 to 119.41] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 14.3
Statistical Analysis 2: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4); [analysis description as in outcome 2, analysis 2]; Test type: Other; Ratios of adjusted geometric means [%] = 106.03, 90% CI 2-sided [95.49 to 117.73] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 15.9

9. Secondary Outcome: Area Under the Concentration-time Curve of Omeprazole in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: The area under the concentration-time curve of omeprazole in plasma over the time interval from 0 to the last quantifiable data point is reported.
  Period 1 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 hours post-dose. Period 2 (Day 2): 15 min pre-dose and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 12 h post-dose. Period 2 (Day 15): 15 min pre-dose, and at 15, 30, 45 min; 1, 1.5, 2, 4, 6, 8, 10, 11, 12 hours post-dose.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Midazolam + Omeprazole (Reference Treatment 2) | Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2) | Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4)
Number analyzed (Participants) | 15 | 13 | 13
h*ng/mL | 287 (78.3) | 304 (72.8) | 267 (61.8)
Statistical Analysis 1: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after a single dose of zongertinib (Test Treatments 2); [analysis description as in outcome 3, analysis 1]; Test type: Other; Ratios of adjusted geometric means [%] = 108.13, 90% CI 2-sided [79.90 to 146.35] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 44.9
Statistical Analysis 2: Comparison: Midazolam + Omeprazole (Reference Treatment 2) vs Midazolam + Omeprazole after multiple doses of zongertinib (Test Treatment 4); [analysis description as in outcome 3, analysis 2]; Test type: Other; Ratios of adjusted geometric means [%] = 97.81, 90% CI 2-sided [75.01 to 127.53] — Ratio calculated as test/reference*100. Intra-individual Geometric coefficient of variation [%] = 38.5

ADVERSE EVENTS:
Time Frame: AE collection timeframe: Repa (R1) & Zonger+Repa (T1, T3): up to 24h; Mida+Ome (R2) & Zonger+Mida+Ome (T2, T4): up to 48h; Zonger: up to 14d post-dose. All-cause mortality: Up to 50 days
Description: Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug.
Groups:
- Repaglinide (Reference Treatment 1): Participants received a single 0.5 mg repaglinide tablet on Day 1 of Period 1, after an overnight fast of at least 10 hours.
- Midazolam + Omeprazole (Reference Treatment 2): Participants received 1 mg midazolam (0.5 mL oral solution) coadministered with a 20 mg omeprazole tablet on Day 2 of Period 1, following an overnight fast of at least 10 hours.
- Zongertinib +Repaglinide (Test Treatment 1): Participants received 120 mg zongertinib (two 60 mg tablets) and a single 0.5 mg repaglinide tablet on Day 1 of Period 2, after an overnight fast of at least 10 hours.
- Zongertinib +Midazolam +Omeprazole (Test Treatment 2): Participants received 120 mg zongertinib (two 60 mg tablets) on Day 1. On Day 2, after one day of zongertinib pretreatment, participants were administered 1 mg, midazolam, coadministered with 20 mg omeprazole, and zongertinib following an overnight fast of at least 10 hours.
- Zongertinib: Participants received 120 mg zongertinib daily (as two 60 mg tablets) from Day 1 to Day 15 of Period 2.
- Zongertinib +Repaglinide (Test Treatment 3): Participants received 0.5 mg repaglinide coadministered with zongertinib on Day 14 of Period 2, after 13 days of zongertinib pretreatment and an overnight fast.
- Zongertinib + Midazolam + Omeprazole (Test Treatment 4): Participants received 1 mg midazolam and 20 mg omeprazole coadministered with zongertinib on Day 15 of Period 2, after 14 days of zongertinib pretreatment and an overnight fast.
Arm/Group | Repaglinide (Reference Treatment 1) | Midazolam + Omeprazole (Reference Treatment 2) | Zongertinib +Repaglinide (Test Treatment 1) | Zongertinib +Midazolam +Omeprazole (Test Treatment 2) | Zongertinib | Zongertinib +Repaglinide (Test Treatment 3) | Zongertinib + Midazolam + Omeprazole (Test Treatment 4)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/16 | 2/16 | 4/16 | 4/14 | 9/14 | 2/14 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Repaglinide (Reference Treatment 1) (N=16) | Midazolam + Omeprazole (Reference Treatment 2) (N=16) | Zongertinib +Repaglinide (Test Treatment 1) (N=16) | Zongertinib +Midazolam +Omeprazole (Test Treatment 2) (N=14) | Zongertinib (N=14) | Zongertinib +Repaglinide (Test Treatment 3) (N=14) | Zongertinib + Midazolam + Omeprazole (Test Treatment 4) (N=14)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT06494761/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT06494761/SAP_001.pdf